CLINICAL TRIAL: NCT01253304
Title: A Single Dose Pharmacokinetic Study of LY2189265 in Subjects With Varying Degrees of Hepatic Impairment
Brief Title: A Single Dose Study of LY2189265 in Subjects With Varying Degrees of Hepatic (Liver) Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13765; H9X-EW-GBDO (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-12-01; First posted 2010-12-03 (Estimated); Results first posted 2014-10-07 (Estimated); Last update posted 2014-10-07 (Estimated); Status verified 2014-10

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dulaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Normal hepatic function (Experimental): LY2189265: A single, subcutaneous (SC) 1.5-milligram (mg) injection on Day 1 in participants with normal hepatic function
  Interventions: Drug: LY2189265
- Mild hepatic impairment (Experimental): LY2189265: A single, SC 1.5-mg injection on Day 1 in participants with mild hepatic impairment (Child-Pugh A)
  Interventions: Drug: LY2189265
- Moderate hepatic impairment (Experimental): LY2189265: A single, SC 1.5-mg injection on Day 1 in participants with moderate hepatic impairment (Child-Pugh B)
  Interventions: Drug: LY2189265
- Severe hepatic impairment (Experimental): LY2189265: A single, SC-1.5 mg injection on Day 1 in participants with severe hepatic impairment (Child-Pugh C)
  Interventions: Drug: LY2189265

INTERVENTIONS:
Drug: LY2189265 — Subcutaneous (SC) injection
  Other Names: Dulaglutide

SUMMARY:
The primary purpose of this study is to help answer the following research questions, and not to provide treatment for any condition:

* To evaluate how much of the study drug (LY2189265) is in the blood of participants with varying degrees of liver impairment compared to those with normal liver function.
* To assess the safety of LY2189265 and any side effects that might be associated with it.

ELIGIBILITY:
Inclusion Criteria:

All Participants (including participants with type 2 diabetes mellitus [T2DM]):

* Male participants - Agree to use a reliable method of birth control (for example, barrier methods) during the study and for at least 3 months following dosing of study drug
* Female participants:

  * Women must be of non-child-bearing potential due to surgical sterilization (hysterectomy, bilateral oophorectomy, or tubal ligation) or menopause
  * Women with an intact uterus are deemed postmenopausal if they are over 45 years old and have had cessation of menses for at least 1 year or have had 6 to 12 months of spontaneous amenorrhea with follicle stimulating hormone (FSH) >40 international units per milliliter (IU/mL) and have not taken hormone replacement therapy or oral contraceptives within 1 year of study start and are otherwise healthy
  * Women who have had cessation of menses for at least 2 years are permitted to take hormone replacement therapy
* Have a body mass index (BMI) between 19.0 and 40.0 kilograms per meters squared (kg/m^2), inclusive, at screening.
* Have venous access sufficient to allow blood sampling
* Are reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures
* Have given written informed consent approved by Lilly and the ethical review board governing the site

Control Participants:

* Overtly healthy participants with normal hepatic function
* Participants with T2DM with normal hepatic function
* Have normal sitting blood pressure and pulse rate as determined by the investigator or with changes compatible with their age and disease status in case of patients with T2DM
* Have clinical laboratory test results within normal reference range for the investigator site or results with minor deviations not considered to be clinically significant by the investigator or with changes compatible with their age and disease status in case of T2DM

Hepatic Impaired Participants:

* Have stable hepatic impairment (such as, post-alcoholic, chronic hepatitis, biliary cirrhosis, or cryptogenic) classified as Child-Pugh Class A, B, or C (mild, moderate, and severe impairment) who are considered by the investigator as acceptable for participation in the study. The hepatic-impaired participant population may include patients with T2DM.
* Have sitting blood pressure and pulse rate compatible with their disease state [including T2DM, if applicable] as determined by the investigator.

Participants with T2DM (All Study Groups)

* Have T2DM controlled with diet and exercise alone or T2DM is stable on a single, oral agent antihyperglycemic medication (metformin, sulfonylureas, repaglinide, nateglinide, acarbose [or other disaccharidase inhibitors], or thiazolidinediones) for at least 3 weeks (3 months for thiazolidinediones) prior to admission
* Have a glycosylated hemoglobin (HbA1C) value at screening (or within 4 weeks prior to screening) of 6.5% to 9.0%
* Have clinical laboratory test results within normal range or deemed clinically insignificant by the investigator. Abnormalities of serum glucose, serum lipids, urinary glucose, and urinary protein consistent with T2DM are acceptable
* Have acceptable blood pressure and pulse rate (sitting), as determined by the investigator

Exclusion Criteria:

All participants (including participants with T2DM)

* Are currently enrolled in, discontinued within the last 30 days from a clinical trial involving use of an investigational drug or device other than the study drug, or are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
* Have known allergies to LY2189265 or related compounds
* Have previously completed or withdrawn from this study or any other study investigating LY2189265
* Have a current, functioning organ transplant
* Show evidence of significant active, uncontrolled, endocrine or autoimmune abnormalities (such as, thyroid disease or pernicious anemia) as judged by the screening physician
* Have shown febrile illness within 3 days prior to screening
* Have an abnormality in the 12-lead electrocardiogram (ECG) that, in the opinion of the investigator, increases the risks associated with participating in the study
* Regularly use known drugs of abuse and/or show positive findings on urinary drug screening that are not otherwise explained by permitted concomitant medications
* Show evidence of human immunodeficiency virus (HIV) and/or positive human HIV antibodies
* Are women with a positive pregnancy test or women who are lactating
* Have donated blood of more than 500 milliliters (mL) within the last month prior to screening
* Have an average weekly alcohol intake that exceeds 21 units per week (men) and 14 units per week (women) (1 unit = 12 ounces [oz] or 360 mL of beer, 5 oz or 150 mL of wine, or 1.5 oz or 45 mL of distilled spirits)
* Are unwilling to stop alcohol consumption for the duration of the study (from screening until the follow-up visit)
* Are participants who smoke more than 10 cigarettes per day, are unwilling to refrain from smoking on the day of LY2189265 administration, or are unable to abide by clinical research unit (CRU) restrictions on other inpatient days
* Have a history or presence of pancreatitis (history of chronic pancreatitis or idiopathic acute pancreatitis) or gastrointestinal disorder, (for example relevant esophageal reflux or gall bladder disease, or any gastrointestinal disease which impacts gastric emptying [such as, gastric bypass surgery, pyloric stenosis, with the exception of appendectomy] or could be aggravated by glucagon like peptide [GLP] analogs). Participants with mild hypertension and dyslipidemia, and participants who had cholecystolithiasis (removal of gall stones) and/or cholecystectomy (removal of gall bladder) in the past, with no further sequelae, may be included in the study at the discretion of the screening physician.
* Are participants deemed to be unsuitable by the investigator for any reason.

Control participants:

* Have a history or presence of cardiovascular (such as, myocardial infarction, cerebrovascular accident, venous thromboembolism), respiratory, renal, endocrine (with exception of participants with T2DM), hematological, neurological disorders, cancer, hepatic (including Gilbert's disease), or dermatological disorders or diseases capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study medication; or of interfering with the interpretation of data
* Show evidence of significant active neuropsychiatric disease
* Have creatinine clearance less than 80 milliliters per minute (mL/min) (as calculated by the Cockcroft-Gault equation)
* Show evidence of hepatitis B and/or positive hepatitis B surface antigen
* Show evidence of hepatitis C and/or positive hepatitis C antibody
* Intend to use:

  * Over-the-counter medication (including herbal remedies/health supplements) within 7 days prior to dosing
  * Prescription medication within 14 days prior to dosing participants with mild, moderate, and severe hepatic impairment
* Show evidence of any significant active disease other than that responsible for or associated with hepatic impairment. Participants with hypertension and hyperlipidemia may be permitted at the investigator's discretion.
* Show, in the opinion of the investigator, evidence of significant neuropsychiatric disease other than Grade 1 hepatic encephalopathy
* Show evidence of spontaneous bacterial peritonitis within 6 months of dosing.
* Show evidence of severe hyponatremia (Sodium [Na] <120 millimoles per liter [mmol/L])
* Show presence of hepatocellular carcinoma
* Have a portal shunt
* Show evidence of severe ascites
* Have hemoglobin <9.0 grams per deciliter (g/dL)
* Have platelet count <40 x 10^9 cells per liter (cells/L)
* Have total serum bilirubin >15 milligrams per deciliter (mg/dL)
* Use medication known to interfere with hepatic metabolism (that is, barbiturates, phenothiazines) or known to alter other major organs or systems

Mild, Hepatic Impaired Participants (Child-Pugh A)

* Show evidence of active renal disease with creatinine clearance <70 mL/min calculated by the Cockcroft-Gault equation.
* Moderate and Severe Hepatic Impaired Subjects (Child-Pugh B and C)
* Show evidence of hepatorenal syndrome as shown by creatinine clearance <50 mL/min calculated by the Cockcroft-Gault equation.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2010-11; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Munich, Germany
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Budapest, Hungary

RESULTS

PARTICIPANT FLOW:
Groups:
- Normal Hepatic Function: LY2189265: A single, subcutaneous (SC), 1.5-milligram (mg) injection on Day 1 in participants with normal hepatic function
- Mild Hepatic Impairment: LY2189265: A single, SC, 1.5-mg injection of LY2189265 on Day 1 in participants with mild hepatic impairment (Child-Pugh A)
- Moderate Hepatic Impairment: LY2189265: A single, SC, 1.5-mg injection of LY2189265 on Day 1 in participants with moderate hepatic impairment (Child-Pugh B)
- Severe Hepatic Impairment: LY2189265: A single, SC, 1.5-mg injection of LY2189265 on Day 1 in participants with severe hepatic impairment (Child-Pugh C)
Period: Overall Study
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Started | 11 | 6 | 6 | 3
Received at Least 1 Dose of Study Drug | 11 | 6 | 6 | 3
Completed | 11 | 6 | 6 | 2
Not Completed | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Participants who received at least one dose of study drug (LY2189265).
Groups:
- Mild Hepatic Impairment: LY2189265: A single, SC, 1.5-mg injection on Day 1 in participants with mild hepatic impairment (Child-Pugh A)
- Moderate Hepatic Impairment: LY2189265: A single, SC, 1.5-mg injection on Day 1 in participants with moderate hepatic impairment (Child-Pugh B)
- Severe Hepatic Impairment: LY2189265: A single, SC, 1.5-mg injection on Day 1 in participants with severe hepatic impairment (Child-Pugh C)
- Total: Total of all reporting groups
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment | Total
Number analyzed (Participants) | 11 | 6 | 6 | 3 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.2 (8.5) | 56.3 (9.2) | 54.3 (4.8) | 64.3 (6.5) | 57.6 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 4 | 1 | 15
  Male | 5 | 2 | 2 | 2 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 10 | 6 | 6 | 3 | 25
  More than one race | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Not Hispanic or Latino | 11 | 6 | 6 | 3 | 26
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Germany | 11 | 6 | 6 | 3 | 26

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics: Maximum Observed Concentration (Cmax)
Description: This measure was calculated using non-compartmental analysis techniques.
Time Frame: Predose to 336 hours postdose
Population: Participants who received at least one dose of study drug (LY2189265) with evaluable concentration data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliter (ng/mL)
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 11 | 6 | 6 | 3
nanograms/milliliter (ng/mL) | 84.5 (29) | 63.0 (30) | 58.1 (28) | 61.3 (18)

2. Primary Outcome: Pharmacokinetics: Time of Maximum Concentration (Tmax)
Description: This measure was calculated using non-compartmental analysis techniques.
Time Frame: Predose to 336 hours postdose
Population: Participants who received at least one dose of study drug (LY2189265) with evaluable LY2189265 concentration data.
Measure: Median (Full Range); unit: hours
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 11 | 6 | 6 | 3
hours | 48.00 [24.02 to 72.02] | 48.01 [47.95 to 72.02] | 59.96 [47.10 to 95.97] | 71.93 [71.90 to 71.98]

3. Primary Outcome: Pharmacokinetics: Area Under the Concentration Versus Time Curve From Time Zero to the Last Quantifiable Concentration (AUC[0-tlast])
Description: This measure was calculated using non-compartmental analysis techniques.
Time Frame: Predose to 336 hours postdose
Population: Participants who received at least one dose of study drug (LY2189265) with evaluable LY2189265 concentration data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms times hour/milliliter(ng*hr/mL
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 11 | 6 | 6 | 3
nanograms times hour/milliliter(ng*hr/mL | 10200 (26) | 7670 (27) | 7220 (19) | 7660 (13)

4. Primary Outcome: Pharmacokinetics: AUC From Time Zero to Infinity (AUC[0-infinity])
Description: This measure was calculated using non-compartmental analysis techniques.
Time Frame: Predose to 336 hours postdose
Population: Participants who received at least one dose of study drug (LY2189265) with evaluable concentration data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms times hr/milliliter (ng*hr/mL)
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 11 | 6 | 5 | 3
nanograms times hr/milliliter (ng*hr/mL) | 16300 (24) | 12200 (26) | 11200 (14) | 12500 (5)

5. Primary Outcome: Pharmacokinetics: Apparent Terminal Elimination Half-life (t1/2)
Description: The half life associated with the terminal rate constant is summarized. This measure was calculated using non-compartmental analysis techniques.
Time Frame: Predose to 336 hours postdose
Population: Participants who received at least one dose of study drug (LY2189265) with evaluable LY2189265 concentration data.
Measure: Geometric Mean (Full Range); unit: hours
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 11 | 6 | 5 | 3
hours | 104 [88.6 to 116] | 101 [86.2 to 116] | 88.2 [75.1 to 104] | 99.2 [76.4 to 121]

6. Primary Outcome: Pharmacokinetics: Apparent Total Plasma Clearance (CL/F)
Description: The apparent total body clearance of drug calculated after extra vascular administration is summarized. This measure was calculated using non-compartmental analysis techniques.
Time Frame: Predose to 336 hours postdose
Population: Participants who received at least one dose of study drug (LY2189265) with evaluable LY2189265 concentration data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters/hour (L/h)
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 11 | 6 | 5 | 3
liters/hour (L/h) | 0.0920 (24) | 0.123 (26) | 0.135 (14) | 0.120 (5)

7. Primary Outcome: Pharmacokinetics: Apparent Volume of Distribution (Vz/F)
Description: The apparent volume of distribution during the terminal phase after extra vascular administration is summarized. This measure was calculated using non-compartmental analysis techniques.
Time Frame: Predose to 336 hours postdose
Population: Participants who received at least one dose of study drug (LY2189265) with evaluable LY2189265 concentration data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters (L)
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 11 | 6 | 5 | 3
liters (L) | 13.8 (27) | 17.9 (27) | 17.1 (20) | 17.1 (24)

ADVERSE EVENTS:
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/6 | 1/6 | 1/3
Other Adverse Events (participants affected / at risk) | 10/11 | 5/6 | 5/6 | 1/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Normal Hepatic Function (N=11) | Mild Hepatic Impairment (N=6) | Moderate Hepatic Impairment (N=6) | Severe Hepatic Impairment (N=3)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Event resulted in death
Peritonitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Status epilepticus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Normal Hepatic Function (N=11) | Mild Hepatic Impairment (N=6) | Moderate Hepatic Impairment (N=6) | Severe Hepatic Impairment (N=3)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Erosive duodenitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eructation (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 2 (6) | 0 (0) | 0 (0)
Reflux oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Varices oesophageal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (3) | 1 (5) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Clostridial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 8 (8) | 4 (4) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral hygroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (3) | 1 (3) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days